CLINICAL TRIAL: NCT05642130
Title: Effect of Muscle Energy Technique on Craniovertebral and Shoulder Angles in Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba saeid Mohamed Ahmed Elfaky, Teaching Assistant, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: P.T.REC/012/003845
Record Dates: First submitted 2022-11-09; First posted 2022-12-08 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2022-11

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Investigator
Masking Description: with computer generated block. Participants were randomized in blocks of 4 with a 1:1 allocation ratio to reduce the bias and variability between the two groups. The randomization was generated by an author who was not entailed in data collection. Randomization codes were kept confidential in sealed opaque envelopes and sequentially numbered to ensure concealed allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental): (30) thirty patients with forward head received PIR for upper trapezius and sternocleidomastoid muscles. the therapist moved the subject's head into the position that put each muscle in stretch, once resistance/ barrier was felt, that position was held and subjects were asked to isometrically contract the target muscle with 20% of maximal contraction for 5 sec against mild resistance from the therapist, relax for 5 sec followed by passive stretch until reaching a new barrier for 30 sec, 3 repetitions for each muscle, 3sessions /week over a period of 4 weeks In addition to the program designed for control group.
  Interventions: Other: exersice program (Muscle energy technique); Other: exersice program (stretching and strengthening exercises ) In addition to postural advices
- control group (Sham Comparator): (30) thirty patients with forward head received static stretching exercise for upper trapezius and sternocleidomastoid .
  Repetitions: 3times/day, 3days/week over a period of 4 weeks, in addition to strengthening exercises of deep cervical flexors and scapular retractor muscles 3sets of 12 repetitions with 6 sec hold. In addition to postural advices
  Interventions: Other: exersice program (stretching and strengthening exercises ) In addition to postural advices

INTERVENTIONS:
Other: exersice program (Muscle energy technique) — Post isometric relaxation for upper trapezius and sternocleidomastoid muscles. the therapist moved the subject's head into the position that put each muscle in stretch, once resistance/ barrier was felt, that position was held and subjects were asked to isometrically contract the target muscle with 20% of maximal contraction for 5 sec against mild resistance from the therapist, relax for 5 sec followed by passive stretch until reaching a new barrier for 30 sec, 3 repetitions for each muscle, 3sessions /week over a period of 4 weeks, In addition to the program designed for control group
  Other Names: post isometricrelaxation for upper trapezius and sternocleidomastoid muscles
  Arms: treatment group
Other: exersice program (stretching and strengthening exercises ) In addition to postural advices — static stretching exercise for upper trapezius and sternocleidomastoid . Repetitions: 3times/day, 3days/week over a period of 4 weeks, in addition to strengthening exercises of deep cervical flexors and scapular retractor muscles, 3sets of 12 repetitions with 6 sec hold. In addition to postural advices
  Other Names: traditional tretment

SUMMARY:
The study will be determine how muscle energy strategy for the upper trapezius and sternocleidomastoid muscles affects the craniovertebral angle and shoulder angle.

DETAILED DESCRIPTION:
Participants in group (A) received PIR for upper trapezius and sternocleidomastoid muscles. the therapist moved the subject's head into the position that put each muscle in stretch, once resistance/ barrier was felt, that position was held and subjects were asked to isometrically contract the target muscle with 20% of maximal contraction for 5 sec against mild resistance from the therapist, relax for 5 sec followed by passive stretch until reaching a new barrier for 30 sec, 3 repetitions for each muscle, 3sessions /week over a period of 4 weeks . In addition to the program designed for control group.

The treatment protocol was designed based on the assumption that the targeted muscles are the most shortened muscles in FHP.

PIR for upper trapezius The patient sat on a stool in an erect position. The therapist stood behind the patient with one hand on the patient's ipsilateral shoulder for stabilization, while the other was on the side of the patient's head. The patient's head was moved to flexion, lateral bending to the opposite side and rotation to the same side of the stretched muscle. The ipsilateral hand pushed the shoulder inferiorly to lengthen the muscle until the restrictive barrier was met, then we asked the patients to raise the shoulder against the hand isometrically then gently stretch the muscle until meeting a new barrier.

PIR for upper trapezius PIR for Sternocleidomastoid The patient sat on a stool in an erect position. The therapist stood behind the patient with her forearm on the patient's ipsilateral shoulder for stabilization, while the hands surrounded the patient's head. The head moved into lateral flexion away from the side of the involvement, rotation to the side of involvement, extension of the lower cervical spine and flexion of upper cervical spine to meet the restrictive barrier. The patient was instructed to push forward against the therapist's hand isometrically, and then gently stretch the muscle until meeting a new barrier.

Group (B) Participants in group (B) received static stretching exercise for upper trapezius and sternocleidomastoid .

Repetitions: 3times/day, 3days/week over a period of 4 weeks, in addition to strengthening exercises of deep cervical flexors and scapular retractor muscles, 3sets of 12 repetitions with 6 sec hold. In addition to postural advices Strengthening of deep cervical flexor muscles Each participant was instructed to sit with his arms relaxed at the side. The area above the lip and under the nose was lightly touched and the patient was asked to tuck his head down and in. The correct movement of tucking the chin in and straightening the spine were verbally reinforced. From sitting position, the patient was asked to tuck chin so that ears were in line with the tip of shoulders.

Strengthening of the scapular retractor muscles The participant sat on a chair without back support. The movement of the medial border of the scapula was gently resisted and the subject pinch them together "retraction". The subject was asked to imagine "holding a quarter between both the shoulder blades". Instructing each subject not to extend the shoulders or elevate the scapulae. The participant then stranded with his hands grasped together behind the lower back (this activity cause scapular adduction). The patient is instructed to adduct scapula and to hold the adducted position with both arms lowered downwards.

Postural education

• Postural advice They were advised that they should not sleep on a foam rubber pillow; should use a chair with proper back support and an arm rest of an appropriate height to provide elbow support while working at a keyboard and computer; should avoid leaning forward toward the screen of a computer or on a desk while writing for a prolonged period; and should avoid prolonged conversation on a telephone while holding the receiver by tilting the neck. Furthermore, the participants were advised to relieve muscle tension after every 20-30 minutes of work by getting up; stretching the arm, shoulder, neck, and back muscles; and walking to turn off the buzzer and reset the timer. They should either avoid prolonged carrying of a bag on any one side of the shoulder or balance the hanging weight of the bag on both sides of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Both sex will be included with age ranged between (18-23) years old
* subject with CVA less than 50°
* subject with shoulder angle less than 52.28°.
* Subjects without neck or shoulder pain or recent shoulder fracture.
* Body mass index between (18-31) Kg/m2
* They will understand and follow instructions included in the test.

Exclusion Criteria:

* Neck pain
* Shoulder pain
* Recent shoulder fracture
* Athlete
* Cervical disc
* Radiculopathy
* Subjects had symptoms of vertigo, dizziness.
* Subjects had visual or auditory problems.
* Subjects had an autoimmune disease or systemic disease

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2023-01-08 (Actual)

PRIMARY OUTCOMES:
craniovertebral angle | one month
  (CVA): It is the angle formed between a horizontal line through the spinous process of C7 and a line from the tragus of the ear It is a measure of forward head posture
shoulder angle | one month
  (SA) : is formed at a line between the center of the humerus and spinous process of C7 and the horizontal line through the center of the humerus. It is a measure of rounded shoulder posture.
Pressure Pain Threshold | one month
  the point at which a non-painful pressure stimulus turns into a painful pressure sensation Subjects' pressure pain thresholds (PPTs) were assessed using a Commander algometer

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

REFERENCES:
- [Background] Andersen LL, Kjaer M, Andersen CH, Hansen PB, Zebis MK, Hansen K, Sjogaard G. Muscle activation during selected strength exercises in women with chronic neck muscle pain. Phys Ther. 2008 Jun;88(6):703-11. doi: 10.2522/ptj.20070304. Epub 2008 Mar 13. PMID 18339796
- [Background] Diab AA, Moustafa IM. The efficacy of forward head correction on nerve root function and pain in cervical spondylotic radiculopathy: a randomized trial. Clin Rehabil. 2012 Apr;26(4):351-61. doi: 10.1177/0269215511419536. Epub 2011 Sep 21. PMID 21937526
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Falla D, Jull G, Russell T, Vicenzino B, Hodges P. Effect of neck exercise on sitting posture in patients with chronic neck pain. Phys Ther. 2007 Apr;87(4):408-17. doi: 10.2522/ptj.20060009. Epub 2007 Mar 6. PMID 17341512
- [Background] Grimmer-Somers K, Milanese S, Louw Q. Measurement of cervical posture in the sagittal plane. J Manipulative Physiol Ther. 2008 Sep;31(7):509-17. doi: 10.1016/j.jmpt.2008.08.005. PMID 18804001